CLINICAL TRIAL: NCT07232745
Title: Mucosal and Systemic Immune Responses Induced by an Intranasal Influenza Live Attenuated Vaccine: A Single-Center, Open-Label, Single-Arm Clinical Study
Brief Title: Mucosal and Systemic Immune Responses Induced by an Intranasal Influenza Live Attenuated Vaccine
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSJKYMS002
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Influenza
Keywords: Systemic Immunity; Mucosal Immunity; Intranasal Influenza Live Attenuated Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The vaccination group (Self-Controlled) (Experimental)
  Interventions: Biological: LAIV

INTERVENTIONS:
Biological: LAIV — This vaccine is produced by Changchun BCHT Biotechnology Co.

SUMMARY:
This is a single-center, open-label, single-arm clinical trial designed to evaluate the mucosal and systemic immune responses induced by an intranasal influenza live attenuated vaccine, and to explore the correlation between the two. The study plans to recruit 60 healthy volunteers aged 14-17 years, with a male-to-female ratio of 1:1. Participants and their guardians must be able and willing to comply with the clinical trial protocol and provide informed consent. Eligible participants will receive a single 0.2 mL dose of LAIV prior to the influenza season. Information on participants' historical vaccination records, baseline demographic data, and past health status will be collected. Nasal specimens (nasal secretions and nasal mucosal cells) and blood samples (serum and PBMCs) will be collected on Day 0 (before vaccination), Day 7, and Day 28 after vaccination for transcriptome sequencing and immunogenicity analysis. In addition, fecal samples will be collected on Day 0 (before vaccination), Day 7, and Day 28 after vaccination for intestinal microbiota detection.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 14-17 years.
2. Volunteers and their guardians are able and willing to comply with the requirements of the clinical trial protocol and sign the informed consent form.

Exclusion Criteria:

1. Allergy to any component of the vaccine product, including eggs, excipients, or gentamicin sulfate.
2. Individuals with acute illnesses, severe chronic illnesses, acute exacerbations of chronic illnesses, or fever.
3. Pregnant or lactating women.
4. Individuals with Leigh syndrome who are receiving treatment with aspirin or aspirin-containing medications.
5. Individuals with immunodeficiency, immunosuppression, or those undergoing immunosuppressive therapy.
6. Individuals with uncontrolled epilepsy, other progressive neurological disorders, or a history of Guillain-Barré syndrome.
7. Individuals with rhinitis or asthma.
8. Individuals with a personal or family history of seizures, chronic diseases, epilepsy, or allergic tendencies.
9. Individuals who have received immunoglobulin injections within the last 3 months prior to vaccination.
10. Individuals who have used other live attenuated vaccines within 1 month prior to vaccination.
11. Individuals planning to use antiviral drugs for influenza within 48 hours before or 2 weeks after vaccination.
12. Individuals planning to use any other intranasal medication within 2 days after vaccination.
13. Subjects with underlying gastrointestinal diseases, including but not limited to inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), chronic diarrhea, peptic ulcer, and intestinal polyps.
14. Subjects with metabolic diseases, such as diabetes mellitus, obesity (BMI ≥ 25.9 kg/m²), hyperlipidemia, or metabolic syndrome.
15. Subjects who have used antibiotics, probiotics, or other drugs that may affect the intestinal microbiota within the past 3 months.
16. Other circumstances in which the subject is deemed unsuitable for participation in the study by the investigator.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
The level of IgG antibodies (ng/mL) against the vaccine strain in serum at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
The level of sIgA antibodies (AU/mL) against the vaccine strain in nasal secretions at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA)

SECONDARY OUTCOMES:
The levels of cytokines in serum at 7 days post-vaccination. | Day 7 post-vaccination
  Measured by Meso Scale Discovery
The levels of cytokines in nasal mucosal secretions at 7 days post-vaccination. | Day 7 post-vaccination
  Measured by Meso Scale Discovery
The levels of cytokines in serum at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Meso Scale Discovery
The levels of cytokines in nasal mucosal secretions at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Meso Scale Discovery
The level of IgG antibodies (ng/mL) against the vaccine strain in serum at 7 days post-vaccination. | Day 7 post-vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA)
The level of neutralizing antibodies (NT50 and IC50, ng/mL) against the vaccine strain in serum at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Neutralization Assay
The gene expression levels in PBMCs (Peripheral Blood Mononuclear Cells) at 7 days post-vaccination. | from baseline (pre-vaccination) to 7 days post-vaccination
  Measured by Bulk Ribonucleic Acid Sequencing.
The gene expression levels in nasal mucosal cells at 7 days post-vaccination. | from baseline (pre-vaccination) to 7 days post-vaccination
  Measured by Bulk Ribonucleic Acid Sequencing.
The gene expression levels in PBMCs (Peripheral Blood Mononuclear Cells) at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Bulk Ribonucleic Acid Sequencing.
The gene expression levels in nasal mucosal cells at 28 days post-vaccination. | Day 28 post-vaccination
  Measured by Bulk Ribonucleic Acid Sequencing.
The level of sIgA antibodies (AU/mL) against the vaccine strain in nasal secretions at 7 days post-vaccination. | Day 7 post-vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA)

OTHER OUTCOMES:
Changes in the abundance of intestinal microbiota compared with baseline (Exploratory). | Day 28 post-vaccination
  Measured by 16s RNA or metagenomic analysis
Changes in the levels of fecal or serum metabolites compared with baseline (Exploratory) | Day 28 post-vaccination
  Ultra-High Performance Liquid Chromatography-Mass Spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Xin Li, PhD, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (1):
- Haizhou District Center for Disease Control and Prevention, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No